CLINICAL TRIAL: NCT05424744
Title: Telemedicine Management of Hypertension: A Pre-Implementation Study
Brief Title: Telemedicine Management of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00085682
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
Keywords: hypertension management; blood pressure monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: enroll up to 10 patients/clinic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine Management of Hypertension (Experimental): using home blood pressure monitoring
  Interventions: Behavioral: Telemedicine Management of Hypertension

INTERVENTIONS:
Behavioral: Telemedicine Management of Hypertension — Telemedicine Management of high blood pressure using home blood pressure monitoring and telemedicine based hypertension self- management support and pharmacotherapy. This will be supplemented by support from community health workers.

SUMMARY:
Explore barriers, facilitators, acceptability, feasibility, and fidelity of the telemedicine management of hypertension intervention

DETAILED DESCRIPTION:
The purpose of the current study is to conduct pre-implementation work to understand the determinants of the telemedicine management of hypertension intervention implementation, feasibility of the intervention and its tailoring, and explore potential inequitable implementation factors in African American patients to enhance the intervention's usability to inform future hybrid trial design.

ELIGIBILITY:
Inclusion Criteria Patients:

* > 18 years of age
* diagnosis of Hypertension (HTN)
* systolic Blood Pressure > 140mmHg on last two clinic visits
* stable anti-HTN medication in the preceding six weeks
* possess smart phone
* must speak and read English

Exclusion Criteria Patients:

* conditions that diminish the ability to conduct home-based self-assessments of Blood Pressure
* chronic conditions that add complexity in HTN management
* recent acute health changes that increases likelihood of Blood Pressure instability
* terminal illness

Inclusion Criteria Stakeholders:

* identify stakeholders using Mendelow's stakeholder matrix, which helps recognize stakeholders according to their interest and power in using the intervention in their clinic - Stakeholders are from clinic and community health workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention (AIM) | Month 3
  Acceptability will be assessed using mixed methods from both patients and stakeholders. The study team will derive themes from relevant constructs about implementation acceptability using qualitative interviews. The study team will complement this using a quantitative measure, Acceptability of Intervention Measure (AIM), which is a validated four item generic implementation outcome measures to assess implementation acceptability. Embedded mixed methods will allow alignment in results of the qualitative and quantitative analyses to provide context, complementarity, and convergence.
Appropriateness of Intervention (IAM) | Month 3
  Appropriateness will be assessed using mixed methods from both patients and stakeholders. The study team will derive themes from relevant constructs about implementation appropriateness using qualitative interviews. The study team will complement this using a quantitative measure, Intervention Appropriateness Measure (IAM), which is a validated four item generic implementation outcome measures to assess implementation appropriateness. Embedded mixed methods will allow alignment in results of the qualitative and quantitative analyses to provide context, complementarity, and convergence.
Feasibility of Intervention (FIM) | Month 3
  Feasibility will be assessed using mixed methods from both patients and stakeholders. The study team will derive themes from relevant constructs about implementation feasibility using qualitative interviews. The study team will complement this using a quantitative measure, Feasibility Intervention Measure (FIM), which is a validated four item generic implementation outcome measures to assess implementation feasibility. Embedded mixed methods will allow alignment in results of the qualitative and quantitative analyses to provide context, complementarity, and convergence. As an additional feasibility outcome, the study team will assess the proportion of eligible and screened patients who agree to participate as well as those who decline (with reasons).
Fidelity of Intervention/implementation | Month 3
  The study team will assess implementation fidelity both at the provider level (number of contacts between patients and nurses; number of pharmacologic activations) and at the patient level (number of home blood pressure data transferred).
Cost Estimates | Month 3
  The study team will estimate cost by calculating the numbers of clinic staff needed and the time spent (by provider type) per patient as well as other resources required for implementation. The study team will document resource commitment (e.g., staff time by provider type [nurses, advanced practice providers, physicians, community health workers], equipment, support [investigative team's support for device set-up, technical and implementation help]) for cost assessments. The study team will stratify cost related to the intervention and implementation strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Yashashwi Pokharel, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manandhar S, Chhetri S, Sutton D, Saha AC, Kaur S, Brown J, Williamson J, Callahan KE, Moore JB, Taylor YJ, Bosworth HB, Pokharel Y. Piloting a team-based telemedicine care for hypertension focused on Black patients. Pilot Feasibility Stud. 2025 Jul 7;11(1):95. doi: 10.1186/s40814-025-01656-y. PMID 40624567

DOCUMENTS (1):
  • Informed Consent Form (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT05424744/ICF_000.pdf